CLINICAL TRIAL: NCT00411866
Title: Open Label Study in Healthy Volunteers to Investigate the Effect of Ketoconazole 400mg on Pharmacokinetics of SB-773812 20mg
Brief Title: Effects Of The Drug Ketoconazole On How The Body Handles The Drug SB773812
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NAA105416
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia
Keywords: safety; pharmacokinetics,
MeSH Terms: conditions — Schizophrenia | interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving ketoconazole for 8 days (Experimental): In Session 1, subjects will receive a single oral dose of SB-773812 20 milligrams (mg), followed by 21 days-washout. In Session 2, subjects will receive once daily oral dose of ketoconazole 400 mg repeated for 8 days. On day 5, single oral dose of SB-773812 20 mg will be dosed concomitantly with ketoconazole.
  Interventions: Drug: SB773812; Drug: Ketoconazole
- Subjects receiving ketoconazole for 14 days (Experimental): In Session 1, subjects will receive a single oral dose of SB-773812 (20mg), followed by 21 days-washout. In Session 2, subjects will receive once daily oral dose of ketoconazole 400 mg repeated for 12 days. On day 5, single oral dose of SB-773812 20 mg will be dosed concomitantly with ketoconazole.
  Interventions: Drug: SB773812; Drug: Ketoconazole

INTERVENTIONS:
Drug: SB773812 — SB-773812 20 mg will be available as white round film coated tablets.
Drug: Ketoconazole — Ketoconazole will be available as 200mg tablets.
  Other Names: SB773812

SUMMARY:
The purposes of this study are to determine if there is a difference in how SB-773812 is distributed through the bloodstream before and after multiple doses of ketoconazole have been given and to determine if there is a difference in how safe and well tolerated SB-773812 is when given on its own and given with ketoconazole.

ELIGIBILITY:
Inclusion criteria:

* Healthy
* Body Weight >/=50kg and BMI 18.5-29.9 kg/m2 inclusive
* Normal 12-lead ECG, physical examination and lab screen

Exclusion criteria:

* A history of psychiatric illness,
* A history or presence gastro-intestinal,
* A hepatic or renal disease or orthostatic hypotension.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10-13 (Actual); Primary Completion 2007-10-10 (Actual); Study Completion 2007-10-10 (Actual)

PRIMARY OUTCOMES:
Blood sampling over period of 336 hours post dosing with SB-773812 | over period of 336 hours post dosing

SECONDARY OUTCOMES:
Safety: ECG, vital signs, adverse events, clinical labs over 48 hours post SB-773812 dosing. | over 48 hours post SB-773812 dosing.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dundee, United Kingdom

REFERENCES:
- See also: Results for study NAA105416 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/NAA105416?search=study&search_terms=NAA105416#rs